CLINICAL TRIAL: NCT01184547
Title: "Effects of a Community Based Exercise Program in Adults With Severe Burns"
Brief Title: Effects of a Community Based Exercise Program in Adults With Severe Burns
Acronym: COMBEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); American Burn Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-034; A-15774.3a (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2010-08-13; First posted 2010-08-19 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Burn Injury; Psychosocial Problem; Quality of Life
MeSH Terms: conditions — Burns | interventions — Return to Work; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COMBEX (Experimental): Community Based Exercise Program or exercise group and quality of life Intervention- The community-based exercise program consisted of 12 weeks of exercise with a community-based trainer after hospital discharge.
  Interventions: Behavioral: Combex
- Standard Of Care (Active Comparator): Standard of Care group, group with no exercise and quality of life. Intervention- No exercise training received.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Combex — 12 weeks of exercise with a trainer post discharge.
  Other Names: Quality of life questionaires-BSHS-B, SF-12, and back to work
  Arms: COMBEX
Behavioral: Standard of Care — No exercise training received.
  Other Names: Quality of life questionaires-BSHS-B, SF-12, and back to work
  Arms: Standard Of Care

SUMMARY:
The purpose of this proposal is to assess the efficacy of implementing a 12-week structured and supervised community-based exercise program (COMBEX) at hospital discharge. The investigators will assess the effect of exercise on mental health and physical function, along with its effects on the amelioration of the burn-induced catabolic response.

The central hypothesis of this proposal is that exercise-induced physical and psychosocial benefits obtained during a supervised and structured COMBEX program in severely burned adults will improve physical function, and quality of life relative to Standard of Care (SOC).

DETAILED DESCRIPTION:
The current Standard of Care in the physical rehabilitation of burned individuals is to discharge them home with prescribed written, physical and occupational therapy rehabilitation activities. We believe that a supervised and structured COMBEX program early during the recovery phase will increase physical function, translate into improvements in QOL, and produce results far superior to current Standard of Care. We intend with this study to eliminate the physical inactivity that occurs with the present standard of care and connect burned victims with COMBEX. This is also important since an inactive lifestyle is a health risk factor even in the physically-able individual. Thus, a fitter burned individual should more readily meet the physical demands of activities of daily living. Activities of daily living, whether occupational or leisure, are integrated functions requiring cardiovascular and muscle endurance and muscle strength. Therefore, successful rehabilitation programs need to also optimize cardiopulmonary and muscle endurance, strength and function; a need that exercise should fulfill. Additionally, a successful rehabilitation program should improve QOL and community engagement. Accordingly, in the present grant application, we propose using exercise as the integral and central interventional tool to counteract physical dysfunction in burned individuals, thereby improving overall functional physical capacity, but also preventing secondary conditions that result from prolonged or maintained physical inactivity and disability. Finally, this increase in physical capacity will allow for an improvement in the QOL of burned individuals, evidenced by increased psychosocial responses measured by increased self-esteem, social interaction, return to work, and decreased anxiety and depression.

We propose to improve the current Standard of Care by the incorporation of a community-based, supervised, structured aerobic and resistive exercise rehabilitation program (COMBEX).

In addition, our present grant proposal attempts to bypass the exercise training in a burn center and translate it into community based facilities. To our knowledge, our studies are the only prospective, randomized studies of exercise and the physiological or psychosocial responses to aerobic or resistance training and quality of life in burned adults.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >18 ≤ 60 years of age and patient agrees to study; 30% Total Body Surface Area (TBSA) burn or greater; AND has been medically cleared for discharge and exercise participation by the treating burn surgeon.

Exclusion Criteria:

* The criteria or risk factors that exclude individuals from this study are:

  * Known history of AIDS, AIDS Related Complex, HIV,
  * Malignant neuroleptic hyperthermia,
  * Active tuberculosis,
  * Arthritis
  * Cirrhosis,
  * Cancer within 5 years
  * Hyperlipidemia
  * Bone or Endocrine Diseases
  * Autoimmune Diseases
  * Chronic Glucocorticoid or non-steroidal anti-inflammatory drug therapy
  * Renal insufficiency (defined by creatinine >3.0 mg/dl),
  * Hepatic disease (defined by elevated liver enzymes or bilirubin >3.0 mg/dl),
  * Known coronary artery disease,
  * Congestive heart failure,
  * Uncontrolled asthma or pulmonary disease (e.g. emphysema, COPD),
  * Associated head injuries requiring specific treatment,
  * Mental retardation or autism or any other mental disorder, which makes it impossible to participate in an exercise program;
  * Gastrointestinal disorders which impair absorption.
  * Pregnancy if applicable

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Burn Specific Health Scale Brief (BSHS-B) | Change from discharge from the ICU to 12 weeks post discharge from ICU.
  The BSHS-B will be used to assess physical functioning and burn injury interference with work activities. The scale for the questionnaire include -0 extremely, 1-Quite a Bit, 2-moderately, 3- a little bit, 4-None (not at All).
Veterans Rand Health Survey 12-item Health Survey (SF-12) | Change from discharge from the ICU to 12 weeks post discharge from ICU.
  The SF-12 is a 12-item; self-report questionnaire that yields two subscales: physical health and mental health.
Return to Work | 12 weeks post discharge from ICU.
  Self-reported, short questionnaire taking approximately 10 minutes to complete. These questionnaires will assess the present employment status and the time from discharge to return to work, past and current employment status as well as job type and, if applicable, start dates for post-injury positions. Time from discharge to return to work will be measured in weeks. The questionnaire ask yes or questions. Also, two scales from 0-10, rate how difficult is to return to work and how satisfied are they are being back to work. 0 is none, 10 is extremely difficult/extremely satisfied.

SECONDARY OUTCOMES:
Peak aerobic capacity | Change from discharge from the ICU to 12 weeks post discharge from ICU.
  A maximal exercise test on a treadmill using the Modified Bruce protocol. VO2peak will be measured by patient's breathing.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar E. Suman, PhD, Principal Investigator — University of Texas/Shriners Hospital for Children
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Voigt CD, Foncerrada G, Pena R, Guillory AN, Andersen CR, Crandall CG, Wolf SE, Herndon DN, Suman OE. Effects of Community-Based Exercise in Adults With Severe Burns: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 Jan;101(1S):S36-S41. doi: 10.1016/j.apmr.2017.12.022. Epub 2018 Jan 31. PMID 29366724